CLINICAL TRIAL: NCT01729962
Title: Comparative Study of the Optical Biometer for the Measurements of Axial Length, Anterior Chamber Depth, Keratometry, Corneal Cylinder Axis, Corneal Thickness, White-to-White Distance, and Pupil Diameter
Brief Title: Comparative Study of the Optical Biometer for Measurements of the Eye
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL-3
Record Dates: First submitted 2012-11-07; First posted 2012-11-21 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Normal Non-fluency; Cataract; Aphakic Eye; Eyes With Corneal Abnormality
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Agreement Cohort: All subjects in the agreement portion of the study will have a single measurement performed with each device, the Nidek optical biometer, predicate device and ultrasound reference device. Each device will be operated by a different operator.
- Precision Cohort: All subjects in the precision portion of the study will each be paired with one Nidek optical biometer and with one predicate device for a total of three Nidek optical biometer/predicate device pairs. Each of the three device pairs will be designated one and only one operator. All subjects in the precision portion of the study will have their measurements repeated three times on each of three Nidek optical biometer and predicate device pairs.

SUMMARY:
The primary purpose of this comparative clinical study is to collect clinical data to demonstrate the equivalence of the investigational device to the predicate device for measurements of the eye. The secondary purpose is to evaluate any adverse events that occur during the clinical study.

DETAILED DESCRIPTION:
This is a prospective clinical study to be conducted at a single clinical site located in the United States. This study will assess the agreement of an investigational device to the predicate device and an ultrasound reference device and the precision of the investigational device with a comparison to the precision of the predicate. Any adverse events associated with the investigational device can or the predicate device will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who can follow the instructions by the Principal/Clinical Investigator or clinical staff at the clinical site, and can visit on scheduled examination dates.
2. Subjects who sign an informed consent form to participate in the clinical trial.
3. Subjects who agree to take the qualifying eye examination and a series of devices measurements.
4. Subjects able to fixate on a target.
5. Subjects must meet at lease one of the following criteria:

   * Normal eyes: Subjects with a natural lens without a cataract, corneal abnormalities or prior keratorefractive surgery.
   * Eyes with Cataracts: Subjects with a pre-existing cataract without corneal abnormalities or prior keratorefractive surgery.
   * Eyes without a Natural Lens: Subjects that are pseudophakic or aphakic without corneal abnormalities or prior keratorefractive surgery.
   * Eyes with Corneal Abnormality: Subjects with a corneal abnormality and a natural lens without a cataract, or Subjects post keratorefractive surgery and a natural lens without a cataract.

Exclusion Criteria:

1. Pregnancy.
2. Any eye condition preventing use of any of the instruments used in the study.
3. Any eye condition which might impair the validity of results from any of the instruments used in the study.
4. Any medical condition, which, in the Investigator's judgment, interferes with the subject's ability to comply with the protocol, compromises subject safety, or interferes with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal eyes(phakic eyes without cataracts or corneal disease), eyes with cataracts, eyes without a natural lens (including aphakic and pseudophakic eyes), eyes with corneal disease (including eyes post keratorefractive surgery).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Agreement and Precision Endpoints Analyses | Subjects will be followed for the duration of the procedure, up to one day.
  The agreement of the Nidek optical biometer with the predicate device will be assessed for the following measures:
  * Axial Length;
  * Keratometry;
  * Corneal Cylinder Axis;
  * Anterior Chamber Depth;
  * Central Corneal Thickness;
  * White-to-White Distance; and
  * Pupil Diameter.
  In addition, the agreement of the Nidek optical biometer with the ultrasound reference device will be assessed for axial length and anterior chamber depth.
  The precision of Nidek optical biometer and the predicate device will be assessed for the following measures:
  * Axial Length;
  * Keratometry;
  * Corneal Cylinder Axis;
  * Anterior Chamber Depth;
  * Central Corneal Thickness;
  * White-to-White Distance; and
  * Pupil Diameter.

SECONDARY OUTCOMES:
Evaluation of Adverse Events Found During the Study | Subjects will be followed for the duration of the procedure, up to one day.
  The safety endpoint is to evaluate any adverse events associated with the Nidek optical biometer or the predicate or reference devices.

OTHER OUTCOMES:
Additional Analyses for the Agreement Portion of the Study | Subjects will be followed for the duration of the procedure, up to one day.
  Additional analyses will examine the intraocular lens (IOL) power calculation from the Nidek optical biometer only based on the subjects enrolled in the agreement portion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Karl G Stonecipher, M.D., Principal Investigator — Physicians Protocol
Locations (1):
- Physicians Protocol, Greensboro, North Carolina, United States